CLINICAL TRIAL: NCT01624220
Title: A Prospective Study Using Implanted Fiducial Markers to Assess Treatment Accuracy and Esophageal Toxicity in Spinal Stereotactic Body Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0190; NCI-2012-01244 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-04

CONDITIONS: Spinal Tumor
Keywords: Spinal tumor; Tumor of the mid or lower spine; Non-small cell lung cancer; Breast cancer; Prostate cancer; Renal cell cancer; Melanoma; Gastrointestinal cancer; Sarcoma; Thyroid cancer; Head and neck primary cancer; Carcinoma of unknown primary; Fiducial markers; Gold seed markers; Spinal stereotactic body radiation therapy; Spinal SBRT; Stereotactic Radiotherapy
MeSH Terms: conditions — Spinal Cord Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell; Melanoma; Gastrointestinal Neoplasms; Sarcoma; Thyroid Neoplasms; Neoplasms, Unknown Primary | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypofractionated Radiation (Experimental): All patients receive CT-guided spinal SBRT using IMRT to maximize conformality of treatment plan to target volume, while sparing normal structures. Dose given to tumor and number of treatments received determined by patient's doctor.
  In second stage, characterize tolerance of esophagus to hypofractionated radiation doses through prospective constraint relaxation and toxicity monitoring. Data collected from Group 1 in first stage will give data on dose delivered to esophagus. Second stage of protocol will begin accrual once Group 1 has filled. Dose constraints used for Groups 3 allow higher dose. Dose constraints for Group 4 represent modest increase of esophageal dose maximums.
  Interventions: Radiation: Spinal SBRT (Higher Dose); Procedure: Gold Seed Implantation; Behavioral: Questionnaires
- ExacTrac Positioning System (Experimental): Analysis performed of ExacTrac positioning system with and without fiducial guidance. Four dimensional CT datasets for simulation will allow use of data from this portion of protocol to characterize degree to which organ at risk (OAR) motion is relevant at each spinal level. 20 patients accrued in two groups of 10, with 10 patients in each rostral-caudal position in the spine (Group 1: T4-T12, Group 2: L1-L5). Imaging done with fiducial markers for this study will not impact patient management. Patients will treated with standard dose constraints to normal tissues.
  Interventions: Radiation: Spinal SBRT (Standard Dose); Procedure: Gold Seed Implantation; Behavioral: Questionnaires

INTERVENTIONS:
Radiation: Spinal SBRT (Standard Dose) — Group 1 and 2: Standard doses of radiation therapy to the normal esophagus while treating the tumor. Up to 2 groups of 10 participants enrolled.
  Other Names: XRT
  Arms: ExacTrac Positioning System
Radiation: Spinal SBRT (Higher Dose) — Group 3 and 4: Higher dose of radiation to esophagus than group before it, if no intolerable side effects were seen. 2 groups of 10 participants enrolled in the second part of study. Only participants who will receive a single spinal SBRT treatment are eligible for second part of study.
  Other Names: XRT
  Arms: Hypofractionated Radiation
Procedure: Gold Seed Implantation — 4 gold seeds implanted into bones of spine: 2 gold seeds above and 2 gold seeds below the area of tumor to be treated.
  Other Names: Fiducial implantation
Behavioral: Questionnaires — Completion of questionnaire before radiation treatment starts, and 1 time a week for the next 4 weeks. It should take about 10 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of the first part of this clinical research study is to learn how to deliver more accurate radiation treatment of tumors in the spine. Researchers also want to learn how internal organs might move during radiation treatment.

The goal of the second part of this study is to learn if it is safe to allow slightly more radiation to the normal esophagus when spinal tumors close by are being treated. This may result in better tumor control.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of 10 participants will be enrolled in the first part of the study, and up to 2 groups of 10 participants will be enrolled in the second part of the study. Only participants who will receive a single spinal SBRT treatment are eligible for the second part of the study.

The participants in the first part of the study will receive standard doses of radiation therapy to normal organs while treating the tumor. In the second part of the study, each new group will receive a higher dose of radiation to the esophagus than the group before it, if no intolerable side effects were seen.

Radiation Planning and Treatment:

Before starting radiation treatment, you will be asked to complete a questionnaire about any symptoms you might be having and any drugs that you are taking. It should take about 10 minutes to complete. After treatment, you will be given copies of the questionnaire to take with you, and asked to fill it out 1 time a week for the next 4 weeks. You should return the questionnaires by mail. Self-addressed stamped envelopes will be given to you.

During all radiation treatments, the images that are taken during your treatment will be closely analyzed after treatment is over. You will have 1 to 3 radiation treatment sessions depending on your doctor's decision.

If you are in the second part of the study, you will receive slightly more radiation than usual to the normal esophagus.

The rest of your radiation treatment planning and treatment delivery appointments will be unchanged. The dose given to the tumor and number of treatments you receive will be determined by your doctor, and is not affected by taking part in this study.

Follow-Up Visits:

After your radiation treatment schedule ends, you will return for follow-up visits at the following time points:

* At 3 months
* Then, every 3 months for 1 year
* Every 6 months during year 2, and then
* 1 time a year after that, for as long as possible

Additional follow up visits may be scheduled, if your doctor thinks they are needed.

At these visits, the following tests and procedures will be performed:

* Any updates to your medical history will be recorded and you will be asked about any side effects you may be having.
* Your performance status will be recorded.
* Your completed symptom questionnaires will be reviewed.
* You will have a physical, including measurement of your vital signs
* You will have a neurological exam.
* You will have follow-up imaging (such as an MRI) to check the status of the disease.

This is an investigational study. Radiation therapy is delivered using FDA-approved and commercially available methods. It is considered investigational to give increased radiation to the esophagus.

Up to 57 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. STAGE 1: >/= 18 years old
2. STAGE 1: Pathologically confirmed diagnosis of cancer, including, but not limited to non-small cell lung cancer, breast, prostate, renal cell, melanoma, gastrointestinal, sarcoma, thyroid, head and neck primary, and carcinoma of unknown primary
3. STAGE 1: Signed informed consent
4. STAGE 2: 1-3 above, and Patients undergoing single fraction spinal SBRT

Exclusion Criteria:

1. STAGE 1: Patient with radiosensitive histologies (lymphoma, multiple myeloma, small cell carcinomas, germ cell tumors)
2. STAGE 1: Extensive (> 50%) height loss of the involved vertebral body
3. STAGE 1: Inability to tolerate lying flat on treatment table for greater than 30 minutes
4. STAGE 1: Pregnancy
5. STAGE 2: Prior irradiation of the spine site and level to be treated
6. STAGE 2: Patients with primary disease arising in the posterior elements of the VB in question
7. STAGE 2: History of Barrett's esophagus, esophageal webbing, stricture, or fistula
8. STAGE 2: Prior radiation to the esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Assess Use of Implanted Fiducial Markers in Treatment Planning and Delivery Workflow for Frame-Based Spinal Stereotactic Body Radiation Therapy (Spinal SBRT) | 1 month
  Establish platform and perform analysis of the ExacTrac positioning system with and without fiducial guidance.
  Patients monitored at each follow-up visit, with MRI of the spine performed at each follow-up time point during the first year. Treated lesions will be classified as progressive (defined as > 25% increased volume), stable (defined as radiographically unchanged), or smaller, and spinal tumor progression-free survival (PFS) will be calculated.

SECONDARY OUTCOMES:
Esophageal Tolerance to Hyperfractionation | 1 month
  Characterize tolerance of esophagus to hypofractionated radiation doses through prospective constraint relaxation and toxicity monitoring.
  Specific esophageal toxicity endpoints monitored include: dyspepsia, dysphagia, fistula, hemorrhage, necrosis, obstruction, pain, perforation, stenosis, ulcer, varices and esophagitis.

CONTACTS AND LOCATIONS:
Overall Officials: Amol J. Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org